CLINICAL TRIAL: NCT03690167
Title: Clinical Investigation of the Effects of Concentrated Growth Factor (CGF) and Advanced Platelet Rich Fibrin (A-PRF) on Pain, Edema and Trismus After Impacted Lower Third Molar Surgery
Brief Title: Investigation of the Effects of CGF and A-PRF on Pain, Edema and Trismus After Impacted Lower Third Molar Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Damla Torul (Other)
Responsible Party: Sponsor-Investigator, Dr. Damla Torul, Research Asistant, Oral and Maxillofacial Surgery, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/163
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Trismus; Edema; Pain; Post-Op Complication
MeSH Terms: conditions — Trismus; Edema; Pain; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concentrated Growth Factor (CGF) (Active Comparator): Participants with impacted lower third molar
  Interventions: Other: Concentrated Growth Factor (CGF)
- Advanced Platelet Rich Fibrin (A-PRF) (Active Comparator): Participants with impacted lower third molar
  Interventions: Other: Advanced Platelet Rich Fibrin (A-PRF)
- Control (Sham Comparator): Participants with impacted lower third molar
  Interventions: Other: Control

INTERVENTIONS:
Other: Concentrated Growth Factor (CGF) — CGF application (9 ml venous blood will harvested from the participants in the CGF group and centrifuged according to the protocol for CGF)
  Arms: Concentrated Growth Factor (CGF)
Other: Advanced Platelet Rich Fibrin (A-PRF) — A-PRF application (9 ml venous blood will harvested from the participants in the CGF group and centrifuged according to the protocol for A-PRF)
  Arms: Advanced Platelet Rich Fibrin (A-PRF)
Other: Control — Nothing applied after extraction
  Arms: Control

SUMMARY:
The objective of this case-control intervention study is to explore the effectiveness of Concentrated Growth Factor (CGF) and Advanced Platelet Rich Fibrin (A-PRF) on Pain, Edema and Trismus After Impacted Lower Third Molar Surgery

DETAILED DESCRIPTION:
In the present study, 75 patient, whose ages ranged between 18-30 and have an impacted lower third molar which is in vertical or mesiyoangular position and has class I and II ramus relationship and class B and C depth, will included. 75 patient will divided randomly into three groups as CGF, A-PRF and Control. After third molar surgery CGF and A-PRF will prepared and applied to the extraction sockets in CGF and A-PRF groups. nothing will applied to the control group. Post operative pain, edema and trismus will measured at 2nd and 7th days.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting asymptomatic impacted lower third molar tooth in the vertical or mesioanguler position according to the Winter classification, Class I and II ramus relation and class B and C depth according to Pell-Gregory classification
* Patients between the ages of 18-30,
* Non-smokers,
* Patients with ASA I status

Exclusion Criteria:

* Who does not want to be volunteer for the study,
* Do not comply with post-operative recommendations,
* Operation lasting more than 30 minutes,
* During pregnancy or lactation,
* Have a chronic systemic disorder that may affect healing.
* Unable to cooperate,
* Post-operative infection,
* Patients with pericoronitis

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Edema-amount change of swelling | Baseline, 2nd and 7th days
  In order to evaluate the amount change of swelling after the operation, horizontal and vertical measurements will be made from 5 reference points including tragus, lip corner, soft tissue pogonion, lateral cantus of the eye and gonion. The first measurement between the tragus-lip corner, the second measurement will be obtained by measuring the horizontal distance between the tragus-soft tissue pogonion. The third measurement will be determined by the measurement of the vertical distance between the outer corner of the eye and the gonion. to determine the change in the swelling measurements performed before surgery and at 2nd-7th days after surgery.

SECONDARY OUTCOMES:
Trismus- degree of change (limitation) in maximum mouth opening | Baseline, 2nd and 7th days
  The maximum mouth opening will be determined as the distance between the right lower and upper right central.
Post operative Pain: visual analog (VAS) scale | 6th and 24th hours, 2nd and 7th days
  For the evaluation of the pain, the visual analog scale (VAS) will be used to express the absence of pain in the initial part on a straight line (0) and the end part to express the unbearable pain (10).
  0 (no pain)--------------------------------------------------------------------------------10 (unbearable pain) Higher values of the scale represent worse outcome.
Post-operative symptom severity (PoSSe) scale | Post operative 7th day
  The evaluation of the change in postoperative quality of life will be done with a scale of post-operative symptom severity (PoSSe) consisting of 15-item questionnaire in which the effect of operation on eating, speech, sensation, appearance, pain, disease and daily activities is evaluated. This questionnaire was divided into subscales corresponding to seven main adverse effects, andfor each possible answer there was a score ranging from 0 to a variable number. For total possible answer there was a score ranging from 0 to a 97.9. Higher values of the scale represent worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Torul, PhD, Study Director — Ordu University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD can share with other researchers on demand